CLINICAL TRIAL: NCT01188980
Title: Detectable Esophageal Early Increase in Blood Supply (EIBS) in Patients With Barrett's Esophagus
Brief Title: Early Increase in Blood Supply in Patients With Barrett's Esophagus
Acronym: EIBS in BE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Herbert C. Wolfsen, Professor of Medicine, Mayo College of Medicine, Director of Endoscopy, Mayo Clinic Florida, Mayo Clinic
Other Study IDs: 09-005328
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (3):
- NoBE (control)
- BE without dysplasia
- BE with dysplasia

SUMMARY:
The purpose of this study is to determine if early Barrett's specialized intestinal metaplasia can be detected by measuring early increased blood supply of the esophageal tissue, with 4 Dimensional Elastic Light-Scattering Fingerprinting, (4D-ELF) technology in real time.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older,
* informed written consent,
* patient scheduled for previously planned upper endoscopy

Exclusion Criteria:

* liver disease;
* gastric antral vascular ectasia (GAVE);any known non-esophageal aerodigestive malignancy;
* severe cardiopulmonary disease precluding endoscopy; presence of conditions not allowing biopsy (e.g. coagulation disorder);
* known familial polyposis syndrome (FAP, HNPCC, Juvenile polyposis, etc.);
* known pregnancy or sexually active females of childbearing age who are not practicing an accepted form of birth control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control Population: Patients with no Barrett's metaplasia scheduled for upper endoscopy at Mayo Clinic Jacksonville.
  Experimental Population: Patients with biopsy-proven Barrett's esophagus and previously scheduled for upper endoscopy at Mayo Clinic Jacksonville.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
determine if early increase blood supply (EIBS)can predict presence of Dysplasia | 10 minutes during standard upper endoscopy
  To determine if early increase blood supply (EIBS), as measured in Barrett's glandular mucosa segment, can predict the presence of Dysplasia in patients with known diagnosis of Barrett's esophagus (BE).

SECONDARY OUTCOMES:
determine if EIBS can predict presence of BE in patients undergoing upper endoscopy | 10 minutes
  EIBS measurements taken from buccal mucosa and esophagus will be compared in patients without BE, patients with BE without dysplasia, and patients with BE dysplasia. EIBS measurements will be obtained from normal squamous mucosa in the mouth, proximal esophagus, areas of BE in the distal esophagus, and measurements from the gastric cardia/hiatal hernia (at least 4 cm below the Z line.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States